CLINICAL TRIAL: NCT02573792
Title: Optical Coherence Tomography for the Etiological Diagnosis of Inflammatory Optic Neuritis
Brief Title: Optical Coherence Tomography and Optic Neuritis (OCTON)
Acronym: OCTON
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RDS_2015_21
Record Dates: First submitted 2015-10-09; First posted 2015-10-12 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Optical Neuritis
Keywords: First onset of optical neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Optic neuritis (ON) can remain isolated or reveal a widespread and chronic disease of the central nervous system (CNS), a multiple sclerosis (MS) or, more rarely, a Devic's neuromyelitis optica (NMO) or a systemic disease.

The optical coherence tomography (OCT) is a retinal imaging technique to measure the thickness of the retina and its different layers with an accuracy of 4-6 µM.

Costello et al have shown that approximately 75% of 54 MS patients have developed within 3 to 6 months after a ON a loss of 10 to 40 µM in the thickness of the peripapillary retinal nerve fiber layer (RNFL).

The etiologic diagnosis of ON has been transformed in recent years. MS can now be diagnosed by McDonald's MRI criteria and NMO by the AQP4 antibodies (anti-aquaporin- 4) antibodies and the anti-MOG (myelin-oligodendrocyte glycoprotein) antibodies.

The diagnosis and prognosis value of the OCT in patients with ON is not well known

ELIGIBILITY:
Inclusion Criteria:

* first onset of an optical neuritis lasting for less than 3 months

Exclusion Criteria:

* Contra-indication to MRI
* Patient opposed to participation in the study
* Pregnant or lactating woman
* Patient under a measure of legal protection
* Absence of affiliation to social security or universal health coverage (CMU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at the Adolphe de Rothschild ophthalmological foundation for the first onset of an optical neuritis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the OCT, expressed as a percentage, for the etiological diagnosis of optical neuritis | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region, France